CLINICAL TRIAL: NCT05295563
Title: Effects of Repeated Botulinum Toxin Injections in Lower Extremity Muscles on Muscle Morphology and Functionality in Children With Cerebral Palsy
Brief Title: Effects of Repeated Botulinum Toxin Injections in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kamile Uzun Akkaya, Principal Investigator, Gazi University
Other Study IDs: KamileUzunAkkaya
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy; Muscle Spasticity; Vascularization
Keywords: Repeated botulinum toxin injections; Muscle morphology; Functionality
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Children who had been injected once or twice before were included in Group 1.
  Interventions: Other: Evaluation
- Group 2: Children who received 3 or more injections were included in Group 2.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Gastrocnemius muscle morphology (cross-sectional area, muscle thickness, fascicle length, pennation angle), muscle stiffness, muscle vascularization and functionality of children with CP will be evaluated.

SUMMARY:
One of the disorders observed in children with cerebral palsy (CP) is abnormal muscle tone, and the most common tone problem is spasticity. Botulinum toxin A (BoNT-A) injections are frequently used to reduce spasticity in CP rehabilitation. BoNT-A injections can be administered as a single dose, and some patients require repeated injections. The aim of this study was to examine the effects of repeated BoNT-A applications applied to the gastrocnemius muscle of children with CP on muscle morphology and functionality.

DETAILED DESCRIPTION:
The study will be planned to include 50 children with CP. The children will be divided into two groups.Children who had been injected once or twice before were included in one group; children who received 3 or more injections were included in the other group.Gastrocnemius muscle morphology (cross-sectional area, muscle thickness, fascicle length, pennation angle) was evaluated by ultrasonography, muscle stiffness was evaluated by shear wave ultrasound elastography, and muscle vascularization was evaluated by Superb Microvascular Imaging method by an experienced radiologist. Functionality of children with CP was evaluated with gross motor function measure (GMFM), time up go test, squat test and vertical jumping tests by an experienced pediatric physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Children with unilateral and bilateral, ambulatory, spastic CP, aged 5-18 years
* Children who had previously been injected with BoNT-A into the gastrocnemius muscle

Exclusion Criteria:

* Children with dyskinetic, ataxic, and hypotonic type CP
* Children with a history of any surgical operation or botulinum toxin injection treatment in the previous 6 months

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with unilateral and bilateral, ambulatory, spastic CP, aged 5-18 years, who had previously been injected with BoNT-A into the gastrocnemius muscle, who can cooperate were included in the study.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Muscle morphology | Through study completion, an average of 1 year
  Gastrocnemius muscle morphology will be evaluated by ultrasonography by an experienced radiologist.
Muscle stiffness | Through study completion, an average of 1 year
  Muscle stiffness will be evaluated by shear wave ultrasound elastography by an experienced radiologist.
Muscle vascularization | Through study completion, an average of 1 year
  Muscle vascularization was evaluated by Superb Microvascular Imaging method by an experienced radiologist.
Functionality 1 | Through study completion, an average of 1 year
  One of the functionality evaluations of children with CP was Gross Motor Funtion Mesaurement (GMFM) by an experienced pediatric physiotherapist.
Functionality 2 | Through study completion, an average of 1 year
  One of the functionality evaluations of children with CP was time up go test by an experienced pediatric physiotherapist.
Functionality 3 | Through study completion, an average of 1 year
  One of the functionality evaluations of children with CP was squat test by an experienced pediatric physiotherapist.
Functionality 4 | Through study completion, an average of 1 year
  One of the functionality evaluations of children with CP was vertical jumping test by an experienced pediatric physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided